CLINICAL TRIAL: NCT00016536
Title: Male Tolerance Study of BufferGel and PRO 2000/5 Gel (P)
Brief Title: Effects of BufferGel and PRO 2000/5 Gel in Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Crossover | Purpose: Prevention
Other Study IDs: HPTN 032; 10693 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2001-05-16; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Antiviral Agents; Mucous Membrane; Spermatocidal Agents; Penis; Epithelium; PRO 2000; Urethra; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: Naphthalene 2-sulfonate polymer
Drug: Carbopol polymer

SUMMARY:
The purpose of this study is to find out if there are any bad effects when BufferGel or PRO 2000/5 Gel are applied to the penis of HIV-infected men.

Microbicides are products to be used by women for placing into the vagina to prevent passing HIV from 1 person to another during sex. Studies have shown 2 investigational microbicides, BufferGel and PRO 2000/5 Gel, to be safe and acceptable for women and HIV-negative men. It is important to see if the side effects of these products are the same in men as those in women and to see if there is any difference in the side effects between circumcised and uncircumcised men.

DETAILED DESCRIPTION:
Topical microbicides are products designed to prevent the sexual transmission of HIV and other disease pathogens. Studies have shown that nonoxynol-9, a detergent microbicide, can cause mucosal erosion and ulceration and increased risk of HIV infection. Attention has been given to developing non-detergent topical microbicides, such as BufferGel and PRO 2000/5 Gel. Studies have shown these products to be safe and acceptable for vaginal use [AS PER AMENDMENT 08/20/01: "however, none of the clinical studies to date have investigated the effects on the penile epithelium and urethral mucosa" has been replaced with: Phase I trials also have been conducted to assess the safety of BufferGel and PRO 2000/5 Gel (P) on the penile epithelium and urethral mucosa. In 1 trial, HIV-uninfected men applied either PRO 2000/5 or a gel containing the inactive ingredients of PRO 2000/5 for 7 days. A few patients reported mild symptoms of genital itching, tingling, irritation, dryness, discoloration, or flaking of the dried gel. In a similar trial comparing BufferGel and K-Y Jelly, a few patients reported similar symptoms.] It is important to determine whether the frequency and severity of adverse events experienced by men is comparable to that observed among women. It is also important to determine whether these adverse events are similar between circumcised and uncircumcised men.

Patients are assigned randomly to 1 of 6 possible sequences of product use. Patients complete 3 weeks of nightly product application (7 consecutive nights each of BufferGel, PRO 2000/5 Gel, and placebo gel) separated by a one-week washout between product-use periods. Patients apply the gel to the shaft and glans of the penis at bedtime, leave on for a minimum of 6 hours, and wash off the next morning. Patients maintain a diary of product application and removal, side effects, and use of other medications. Follow-up evaluations, including a genital exam and urine testing, are performed after each product-use and washout period. [AS PER AMENDMENT 08/20/01: Digital photographs will be taken of any observed abnormality or normal area that is needed for clinical decision making and/or documentation purposes.] In addition, adherence is assessed, the patient diary is reviewed, and product acceptability questionnaires are administered after each product-use period. Patients receive monetary compensation for participation.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are male and at least 18 years old.
* Are HIV-positive.
* Have a CD4 cell count over 200 within the year before study entry.
* Can speak and write English.
* Can provide address, phone number, or other contact information.
* Agree not to apply other products to the penis during the 3 weeks of product use.
* Agree not to have sex, masturbate, or perform other activities that may irritate the penis during the 3 weeks of product use.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are allergic to any ingredients in the study products.
* Have had inflammation of the urethra (painful urination, burning, or itching) in the past.
* Have had penis skin reactions, eczema, psoriasis, severe seborrheic dermatitis, or other similar problems in the past.
* Have had a non-HIV sexually transmitted disease (STD), including a genital herpes outbreak, in the past 6 months.
* Have had a change in anti-HIV drugs in the past 30 days.
* Have taken part in any other study of an investigational product in the past 30 days.
* Have broken skin on the penis.
* Have signs or symptoms of an STD.
* Apply topical products (e.g., creams or ointments) to the penis.
* Have an abnormal finding on the physical or genital exam.
* Have a positive result from a urine leukocyte esterase (LE) test.
* Use any drugs that would affect the study, in the doctor's opinion.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Study Completion 1997-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum, Study Chair
Locations (1):
- UW HIV Prevention CRS, Seattle, Washington, United States

REFERENCES:
- [Result] Tabet SR, Callahan MM, Mauck CK, Gai F, Coletti AS, Profy AT, Moench TR, Soto-Torres LE, Poindexter III AN, Frezieres RG, Walsh TL, Kelly CW, Richardson BA, Van Damme L, Celum CL. Safety and acceptability of penile application of 2 candidate topical microbicides: BufferGel and PRO 2000 Gel: 3 randomized trials in healthy low-risk men and HIV-positive men. J Acquir Immune Defic Syndr. 2003 Aug 1;33(4):476-83. doi: 10.1097/00126334-200308010-00008. PMID 12869836